CLINICAL TRIAL: NCT00098969
Title: Phase I Single-Dose Safety and Phamacokinetics Clinical Study of Resveratrol AKA IRB 2003-424
Brief Title: UMCC 2003-064 Resveratrol in Preventing Cancer in Healthy Participants
Acronym: IRB 2004-535
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Prevention
Other Study IDs: CDR0000396464; P30CA046592 (NIH); CCUM-2004-0535; CCUM-2062
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2010-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Resveratrol

INTERVENTIONS:
Drug: resveratrol

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of resveratrol may prevent cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of resveratrol in preventing cancer in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the concentration of resveratrol and its metabolites in the plasma, urine, and feces of healthy participants.
* Correlate dose with systemic concentration of this drug and its metabolites in these participants.
* Determine the safety of this drug in these participants.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Beginning 5 days before study drug administration, participants are put on a controlled diet (avoiding all resveratrol-containing food or drink) for washout. Participants receive oral resveratrol once on day 1.

Cohorts of 10 participants receive escalating doses of resveratrol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 10 participants experience dose-limiting toxicity. A total of 16 participants are treated at the MTD.

Participants are followed at 2 and 7 days.

PROJECTED ACCRUAL: A total of 10-40 participants will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count 120,000-450,000mm^3
* Hemoglobin 10.5-17.5 g/dL for women OR 11.5-19.0 g/dL for men

Hepatic

* Bilirubin 0.05-1.2 mg/dL
* AST and ALT < 1.5 times normal

Renal

* Creatinine normal
* Urinalysis normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective contraception
* Willing to abstain from ingesting large quantities of resveratrol-containing foods
* Willing to spend 24 hours in the hospital
* No cancer diagnosis that is currently under treatment, is clinically detectable, or that has been treated within the past 5 years except basal cell or squamous cell skin cancer
* No concurrent excessive alcohol intake (>21 units per week for men; 14 units per week for women)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent hormone replace ment therapy allowed
* Concurrent oral or depot contraceptives allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 2 weeks since prior and no concurrent vitamin supplements of any type
* More than 6 months since prior and no concurrent participation in any other experimental study
* No other concurrent chronic medications, including over-the-counter medications, herbal/natural preparations, or dietary supplements
* No other concurrent prescribed medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Dean E. Brenner, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States
- Leicester Royal Infirmary, Leicester, England, United Kingdom

REFERENCES:
- [Result] Boocock DJ, Gescher AJ, Brown V, et al.: Phase I single-dose safety and pharmacokinetics clinical study of the potential cancer chemopreventive agent resveratrol. [Abstract] American Association for Cancer Research: 97th Annual Meeting, April 1-5, 2006, Washington, DC. 2006.
- [Derived] Brown VA, Patel KR, Viskaduraki M, Crowell JA, Perloff M, Booth TD, Vasilinin G, Sen A, Schinas AM, Piccirilli G, Brown K, Steward WP, Gescher AJ, Brenner DE. Repeat dose study of the cancer chemopreventive agent resveratrol in healthy volunteers: safety, pharmacokinetics, and effect on the insulin-like growth factor axis. Cancer Res. 2010 Nov 15;70(22):9003-11. doi: 10.1158/0008-5472.CAN-10-2364. Epub 2010 Oct 8. PMID 20935227